CLINICAL TRIAL: NCT01964781
Title: The Effect of Topical Administration of Tranexamic Acid, Adrenaline and Bupivacain on Postoperative Bleeding and Pain in Patients Undergoing Breast Surgery. A Four-armed Placebo-controlled Double Blinded Randomized Study
Brief Title: The Effect of Topical Administration of Common Drugs on Postoperative Bleeding and Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012-004964-23; 2012-004964-23 (EudraCT Number)
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Pain, Postoperative; Postoperative Hemorrhage
Keywords: Administration, topical; tranexamic acid; adrenaline; bupivacaine; surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Hemorrhage | interventions — Tranexamic Acid; Bupivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- topical tranexamic acid (Experimental): tranexamic acid to be smeared on surgical wounds before closure
  Interventions: Drug: Tranexamic Acid
- topical adrenaline (Experimental): adrenaline solution to be smeared on surgical wounds before closure
  Interventions: Drug: Adrenaline
- topical bupivacaine (Experimental): bupivacaine to be smeared on surgical wounds before closure
  Interventions: Drug: Bupivacaine
- topical adrenaline plus tranexamic acid (Experimental): tranexamic acid and adrenaline to be smeared on surgical wounds before closure
  Interventions: Drug: Tranexamic Acid; Drug: Adrenaline
- placebo control (Placebo Comparator): saline to be smeared on surgical wounds before closure
  Interventions: Drug: saline
- tranexamic acid and placebo control (Placebo Comparator): tranexamic acid and saline to be smeared on surgical wounds before closure
  Interventions: Drug: tranexamic acid plus saline

INTERVENTIONS:
Drug: Tranexamic Acid — Topical administration - does it reduce surgical bleeding?
  Arms: topical adrenaline plus tranexamic acid; topical tranexamic acid
Drug: Bupivacaine — Topical Bupivacaine- does it reduce surgical pain?
  Other Names: Marcaine
  Arms: topical bupivacaine
Drug: Adrenaline — Topical adrenaline - does it reduce bleeding on its own, and does it enhance the effect of tranexamic acid?
  Arms: topical adrenaline; topical adrenaline plus tranexamic acid
Drug: tranexamic acid plus saline
  Arms: tranexamic acid and placebo control
Drug: saline
  Arms: placebo control

SUMMARY:
After surgical procedures, interventions to reduce postoperative pain and bleeding are of great importance. In this study, the effect will be investigated of smearing common drugs, which are designed for injection, directly onto the raw wound surface (topical application) created during surgery. Topical application allows a small amount of drug to reach a large wound area, higher drug concentration in the exposed wound surface but very low concentration in the body, and no risk of injury from needles. Although beneficial effects of such an easy and low-cost intervention would be expected, the investigators have found no previous reports on blinded and controlled studies.

DETAILED DESCRIPTION:
The drugs to be studied on whether they reduce bleeding are adrenaline (constricts blood vessels) and tranexamic acid (TXA) (prevents bloodclots from dissolving). The drug studied to what extent it reduces pain will be bupivacaine, a common local anaesthetic. Patients undergoing bilateral symmetric breast surgery or single sided mastectomies are candidates for enrollment in the study. The bilateral patients will have two identical procedures and hence two identical wounds in the same patient. This enables the investigators to use one side as control and hence design our study arms as prospective and placebo-controlled. The patients undergoing a one-sided procedure will need to be compared to similar patients, but as wounds will be of different sizes and in different people, larger groups are needed to find significant differences between treatment and controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral simple mastectomy
* patients undergoing bilateral symmetric breast surgery

Exclusion Criteria:

* pregnancy
* A history of former thromboembolic events (to receive TXA)
* cardiovascular disease (to receive adrenaline)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Amount of blood on drains postoperatively | 24 hours postoperatively
  Drains are placed in surgical wounds during operation, and amount of blood on drains measured in ml on the control after 24 hours.
Amount of pain in operated breast | Measured 24 hours postoperatively
  Evaluate using a visual analogue scale the pain in the surgical wounds as reported by the patient 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Pleym, MD PhD, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843